CLINICAL TRIAL: NCT03597646
Title: The Effect of Kinesio Taping Method and Breathing Exercises on Pulmonary Function, Respiratory Muscle Strength, Functional Capacity and Quality of Life in Patients With Chronic Heart Failure
Brief Title: The Effect of Kinesio Taping on Pulmonary Function and Functional Capacity in Patients With Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Kinesio Taping Association International (Unknown)
Responsible Party: Principal Investigator, Baha Naci, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-29
Record Dates: First submitted 2018-07-01; First posted 2018-07-24 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Chronic Heart Failure
Keywords: Kinesio Taping; inspiratory muscle training; respiratory
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Kinesio Taping (Experimental): Kinesio Taping group consisted of 19 patients. Kinesio Tape was applied 2 times a week for a period of 4 weeks. Kinesio Taping was applied for musculus diaphragmaticus, musculus externus obliquus abdominis and internus obliquus abdominis.
  Interventions: Device: Kinesio Tape
- Inspiratory Muscle Training (IMT) (Active Comparator): Inspiratory Muscle Training (IMT) group consisted of 19 patients. IMT sessions were applied 2 sessions/everyday for a period of 4 weeks and 15 minutes for each session. Every session patients performed 5 breathing circles, then rested and continued again. By this way they used the device for 15 minutes each session. The patients visited the clinic every week and the therapist adjusted the IMT device in terms of their maximal inspiratory pressures.
  Interventions: Device: Threshold Inspiratory Muscle Trainer
- Control (No Intervention): Control group also consisted of 19 CHF patients. No interventions were applied for them. Pharmacological treatment of control group continued and they were advised for using their medication properly.

INTERVENTIONS:
Device: Kinesio Tape
  Other Names: Medical Adhesive Tape
  Arms: Kinesio Taping
Device: Threshold Inspiratory Muscle Trainer
  Arms: Inspiratory Muscle Training (IMT)

SUMMARY:
This randomised controlled study investigates the effect of Kinesio Taping on pulmonary function, respiratory muscle strength, functional capacity, functional mobility, hand grip strength, quality of life and level of depression in patients with chronic heart failure (CHF). The study also compares effects of Kinesio Taping and Inspiratory Muscle Training (IMT). There were 3 study groups: The experimental group received Kinesio Taping; the breathing exercise group received IMT; and the control group received no interventions.

DETAILED DESCRIPTION:
Individuals with chronic heart failure (CHF) have been found to have poor respiratory muscle strength and endurance. The reduction of respiratory muscle strength may be a sign of increased work of breathing in CHF. Exercise intolerance and dyspnea are common symptoms of patients with CHF and are relevant with a poor functional capacity and quality of life. The primary aim of cardiac rehabilitation programs for CHF patients is to increase their exercise tolerance and quality of life. Patients with CHF have decreased lung volume, increased work of breathing, and greater oxygen consumption. Pulmonary rehabilitation may improve quality of life and exercise capacity in patients with CHF. It has been shown that inspiratory muscle training is beneficial for improving respiratory muscle strength, functional capacity, and dyspnea in patients with stable heart failure and respiratory muscle weakness.

It has been found that inspiratory muscle training (IMT) results in improvement in inspiratory muscle strength, functional capacity and quality of life of patients with CHF and inspiratory muscle weakness. Previous studies have shown that the diaphragm has circulatory functions in addition to its better known respiratory functions, that diaphragm strength and endurance diminish in CHF.

Kinesio taping is a relatively new bandaging technique usually applied to normalize muscle function, increase lymph and blood circulation, decrease pain and/or aid the correction of joint misalignment. In literature there are several studies demonstrating results of inspiratory muscle training on pulmonary function in patients with CHF. But we haven't found any studies demonstrating effects of kinesio taping on respiratory mechanics and exercise capacity in patients with CHF. The study we designed therefore may contribute to the literature and may inform future studies.We hypothesized that KT methods used for respiratory muscles would be effective on improving pulmonary function, respiratory muscle strength, quality of life, functional capacity of CHF patients.

Clinically stable 57 CHF patients with New York Heart Association (NYHA) functional class II-III, between the ages 43 and 89 participated in the study. All participants were recruited between September 2016 and February 2017. All the assessments and treatments were performed in the same hospital, Istanbul University Institution of Cardiology, by the same person. The experimental group received Kinesio Taping; the breathing exercise group received IMT; and the control group received no interventions. The Kinesio Taping group received KT facilitation technique for musculus diaphragmaticus (ventral and dorsal parts) and for musculus obliquus internus-externus abdominis (bilateral) to improve inspiratory and forced expiratory muscle activity, respectively. KT was applied twice a week during a 4-week period. By combination of these muscle techniques we investigated the changes in pulmonary functions, respiratory muscle strength, functional exercise capacity, functional mobility, hand grip strength, quality of life and level of depression. All the assessments were performed at baseline and four weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Diagnosed with New York Heart Association Functional Class II-III
* Ejection fraction less than 50
* Stable Chronic Heart Failure patients

Exclusion Criteria:

* Acute decompensated heart failure
* Uncontrolled hypertension
* Unstable angina
* Significant cardiac arrhythmias
* Severe cognitive impairment

Ages: 43 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2017-02-10 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity | 4 weeks
  Forced vital capacity [FVC] (L) was measured with a lung spirometry. This shows the amount of air that the patient can forcefully exhale. The patient sitting on a chair used a nose clips during the test. The patient was asked to take a deep breath from a mouthpiece and then was asked a full forced exhalation for at least 6 seconds. 3 repetitions were performed for each test and best score was accepted.
Forced expiratory volume in 1 second | 4 weeks
  Forced expiratory volume in 1 second [FEV1] (L) was measured with a lung spirometry as it was described for FVC measurement. It shows the amount of air that the patient can forcefully exhale in one second of the FVC test.
FEV1/FVC | 4 weeks
  FEV1/FVC (%) ratio is a very important parameter to determine whether the type of lung disease is obstructive or restrictive.
Peak expiratory flow | 4 weeks
  Peak expiratory flow [PEF] (L/sec) was measured with a lung spirometry as it was described for FVC and FEV1 measurements.
Forced expiratory flow at 25-75% of FVC | 4 weeks
  Forced expiratory flow at 25-75% of FVC [FEF25-75] (L/sec) was measured with a lung spirometry as it was described for FVC, FEV1 and PEF measurements.
Maximal inspiratory pressure | 4 weeks
  Maximal inspiratory pressure [MIP] (cmH2O) was recorded by using a portable mouth pressure meter as a measure of the inspiratory muscle strength. The patient sat upright and took a deep breath from functional residual capacity through a mouthpiece. 5 repetitions repetitions were performed for the test.
Maximal expiratory pressure | 4 weeks
  Maximal expiratory pressures [MEP] (cmH2O) was recorded by using a portable mouth pressure meter as a measure of the expiratory muscle strength. The patient performed a forced expiration from total lung capacity. 5 repetitions repetitions were performed for the test.
Six-minute walk test | 4 weeks
  Functional capacity was determined with Six-minute walk test [6MWT] (m). 6MWT is a submaximal exercise test. For the test we used a 30-m corridor and measured the distance walked by the patient in 6 minutes. We instructed the patient to walk as far as possible. Higher distance indicate better functional capacity.
Short Form-36 | 4 weeks
  Short Form-36 [SF-36] (0-100) was performed to assess generic quality of life (QOL) SF-36 consists of 36 items and 8 subscales. These subscales are physical functioning, role functioning physical, bodily pain, general health perception, vitality, social functioning, role functioning emotional, and mental health and they range from 0 to 100. Higher scores indicate better quality of life.
Minnesota Living with Heart Failure Questionnaire | 4 weeks
  Minnesota Living with Heart Failure Questionnaire [MLHFQ] (0-105) was performed to assess disease-specific QOL.
  MLHFQ consists of 21 items with a total score of 105. Item-level scores of MLHFQ range from 0-5. 8 questions are related to physical domain and 5 questions are related to emotional domains. Total score was calculated by summing all scores. Lower scores indicate better quality of life.

SECONDARY OUTCOMES:
Level of Depression | 4 weeks
  Measured with Beck Depression Inventory. This is a 21-item scale and each question has four possible answers with a score of 0 to 3, and a total score of 0 to 63. A score of 10 or above indicates depression.
Handgrip strength | 4 weeks
  Handgrip strength (kg) was measured by using a hand dynamometer. Patient held the dynamometer in the hand which would be tested. Then the patient squeezed the device with maximum effort in standing position. Then the subject performed this test with the other hand. 3 repetitions were performed for both hands.
Timed up and go test | 4 weeks
  Functional mobility was measured with Timed up and go test [TUGT] (sec). The patient sitting on chair stood up with the instruction of physiotherapist and walked 3 meters as fast as possible, walked back to the chair and sat down again. The total duration was recorded in seconds. Lower time reflects better functional mobility. TUGT was performed with 3 repetitions.
Sit to Stand Test | 4 weeks
  Sit to Stand Test [STS test] (repetitions in 30 seconds) was also used to measure functional mobility. Patient sitting on a 48 cm height armless chair folded their arms across their chests. They stood up completely and then sat down with full contact for a period of 30 seconds. Standing up and sitting down on the chair is one cycle. We calculated the total cycle the patient performed in 30 seconds. Higher score indicates better functional mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Baha Naci, MsC, Principal Investigator — Istanbul University Institution of Cardiology, Istanbul, Turkey; Rengin Demir, Prof., Study Director — Istanbul University Institution of Cardiology, Istanbul, Turkey
Locations (1):
- Istanbul University Institution of Cardiology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McParland C, Krishnan B, Wang Y, Gallagher CG. Inspiratory muscle weakness and dyspnea in chronic heart failure. Am Rev Respir Dis. 1992 Aug;146(2):467-72. doi: 10.1164/ajrccm/146.2.467. PMID 1489142
- [Background] Aubier M, Trippenbach T, Roussos C. Respiratory muscle fatigue during cardiogenic shock. J Appl Physiol Respir Environ Exerc Physiol. 1981 Aug;51(2):499-508. doi: 10.1152/jappl.1981.51.2.499. PMID 6790504
- [Background] Mancini DM, Henson D, LaManca J, Levine S. Respiratory muscle function and dyspnea in patients with chronic congestive heart failure. Circulation. 1992 Sep;86(3):909-18. doi: 10.1161/01.cir.86.3.909. PMID 1516204
- [Background] Adamopoulos S, Schmid JP, Dendale P, Poerschke D, Hansen D, Dritsas A, Kouloubinis A, Alders T, Gkouziouta A, Reyckers I, Vartela V, Plessas N, Doulaptsis C, Saner H, Laoutaris ID. Combined aerobic/inspiratory muscle training vs. aerobic training in patients with chronic heart failure: The Vent-HeFT trial: a European prospective multicentre randomized trial. Eur J Heart Fail. 2014 May;16(5):574-82. doi: 10.1002/ejhf.70. Epub 2014 Mar 14. PMID 24634346
- [Background] Figueroa MS, Peters JI. Congestive heart failure: Diagnosis, pathophysiology, therapy, and implications for respiratory care. Respir Care. 2006 Apr;51(4):403-12. PMID 16563194
- [Background] Lin SJ, McElfresh J, Hall B, Bloom R, Farrell K. Inspiratory muscle training in patients with heart failure: a systematic review. Cardiopulm Phys Ther J. 2012 Sep;23(3):29-36. PMID 22993500
- [Background] Dall'Ago P, Chiappa GR, Guths H, Stein R, Ribeiro JP. Inspiratory muscle training in patients with heart failure and inspiratory muscle weakness: a randomized trial. J Am Coll Cardiol. 2006 Feb 21;47(4):757-63. doi: 10.1016/j.jacc.2005.09.052. Epub 2006 Jan 26. PMID 16487841
- [Background] Mancini DM, Henson D, La Manca J, Donchez L, Levine S. Benefit of selective respiratory muscle training on exercise capacity in patients with chronic congestive heart failure. Circulation. 1995 Jan 15;91(2):320-9. doi: 10.1161/01.cir.91.2.320. PMID 7805234
- [Background] Laoutaris I, Dritsas A, Brown MD, Manginas A, Alivizatos PA, Cokkinos DV. Inspiratory muscle training using an incremental endurance test alleviates dyspnea and improves functional status in patients with chronic heart failure. Eur J Cardiovasc Prev Rehabil. 2004 Dec;11(6):489-96. doi: 10.1097/01.hjr.0000152242.51327.63. PMID 15580060
- [Background] Beeler R, Schoenenberger AW, Bauer P, Kobza R, Bergner M, Mueller X, Schlaepfer R, Zuber M, Erne S, Erne P. Improvement of cardiac function with device-based diaphragmatic stimulation in chronic heart failure patients: the randomized, open-label, crossover Epiphrenic II Pilot Trial. Eur J Heart Fail. 2014 Mar;16(3):342-9. doi: 10.1002/ejhf.20. Epub 2013 Dec 6. PMID 24464736